CLINICAL TRIAL: NCT05447962
Title: Community-engaged Implementation Study of Hypertension Prevention and Navigation in Black Men
Brief Title: Community-engaged Hypertension Prevention Program in Black Men
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-01586
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Barbershop-based facilitation; Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barbershop-Based Facilitation (BF) (Experimental): Participants will receive the Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP) program manual and receive exposure to Barbershop-Based Facilitation (BF), which is designed to stimulate specific, actionable steps that community health workers (CHWs) can undertake to implement CLIP at the barbershop.
  Interventions: Behavioral: Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP); Behavioral: Barbershop-Based Facilitation (BF)
- Self-Directed (Active Comparator): Participants will receive the Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP) program manual.
  Interventions: Behavioral: Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP)

INTERVENTIONS:
Behavioral: Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP) — Multilevel intervention designed to mitigate adverse social determinants of health (SDoH) via linkage to care, health system navigation, and referral to social services.
Behavioral: Barbershop-Based Facilitation (BF) — Trained and qualified facilitators assist community health workers (CHWs) to: 1) increase their confidence in delivering CLIP; 2) understand participants' concerns and beliefs about hypertension (HTN); and 3) develop skills in lifestyle counseling to help the men initiate lifestyle modification.
  Arms: Barbershop-Based Facilitation (BF)

SUMMARY:
The CLIP program will train Community Health Workers (CHWs) to screen and identify Black men with elevated blood pressure (BP) or stage 1 hypertension (HTN), initiate lifestyle counseling; and link them to primary care and social services.

DETAILED DESCRIPTION:
The study will consist of:

1. An implementation phase that will use a cluster randomized cluster trial of 20 barbershops among Black men with elevated BP or Stage 1 HTN, to compare the effect of the Barbershop-based Facilitation (BF) strategy (n=10 barbershops; n=210 participants) vs. self-directed control (i.e. receipt of information for implementation of CLIP without the BF strategy; n=10 barbershops; n=210 participants), on BP reduction, HTN prevention, linkage to care, and adoption of CLIP at 12 months
2. A post-implementation phase that will use Reach Effectiveness Adoption Implementation and Maintenance (RE-AIM) to evaluate the effect of the BF strategy versus self-directed control on sustainability of CLIP 6 months after completion of the trial; and cost-effectiveness over a 10-year time horizon.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age as of date of data extraction
2. Repeat customer within the last 3 months
3. Self-identify as Black
4. Self-identify as male
5. Have elevated blood pressure (PB) (120-129/<80 millimeters of mercury (mm Hg)) or untreated stage 1 hypertension (HTN) (130-139/80-89 mm Hg) (defined by American Heart Association's 2017 HTN clinical guidelines)

Exclusion Criteria:

1. Age <18 years
2. Prescribed antihypertensive medication
3. Diagnosis of end-stage renal disease (ESRD)
4. Condition which interferes with outcome measurement (e.g., dialysis)
5. Serious medical condition which either limits life expectancy or requires active management (e.g., cancer)
6. Cognitive impairment or other condition preventing participation in the intervention
7. Upper arm circumference >50 cm (maximum limit of the extra-large BP cuff)
8. Active alcohol or substance use disorder (i.e., not sober/abstinent for ≥ 30 days)
9. Pregnant or planning pregnancy in the next 24 months
10. Currently nursing a child
11. Current participation in another research study focused on reducing BP
12. Unwillingness to provide informed consent

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-identification.
Enrollment: 430 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) Levels | Baseline, Month 12
  All participants will have office blood pressure (BP) measured on their non-dominant arm with an Omron HEM-907XL BP device.
  3 BP readings separated by one minute will be obtained at each visit. The 3 BP readings will be averaged to obtain mean BP.
  SBP Levels are classified as follows:
  * Normal: Below 120 millimeters of mercury (mm Hg)
  * Elevated: 120-129 mm Hg
  * Stage 1 hypertension: 130-139 mm Hg
  * Stage 2 hypertension: 140 mm Hg or more
  * Hypertensive crisis: 180 mm Hg or more

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure (DBP) Levels | Baseline, Month 12
  All participants will have office blood pressure (BP) measured on their non-dominant arm with an Omron HEM-907XL BP device.
  At each visit, 3 BP readings separated by one minute will be obtained. The 3 BP readings will be averaged to obtain study BP.
  DBP Levels are classified as follows:
  * Normal: Lower than 80 millimeters of mercury (mm Hg)
  * Stage 1 hypertension: 80-89 mm Hg
  * Stage 2 hypertension: 90 mm Hg or more
  * Hypertensive crisis: 120 mm Hg or more.
Number of Participants Presenting to Referral Clinics within 3 Months of Community Health Worker (CHW) Referral | Baseline
  Measurement of linkage to care. Data will be gathered via telephone interview or during barbershop visit.
Number of Participants Presenting to Referral Clinics within 3 Months of Community Health Worker (CHW) Referral | Month 6
  Measurement of linkage to care. Data will be gathered via telephone interview or during barbershop visit.
Number of Participants Presenting to Referral Clinics within 3 Months of Community Health Worker (CHW) Referral | Month 12
  Measurement of linkage to care. Data will be gathered via telephone interview or during barbershop visit.
Number of Participants Presenting to Referral Clinics within 3 Months of Community Health Worker (CHW) Referral | Month 18
  Measurement of linkage to care. Data will be gathered via telephone interview or during barbershop visit.
Number of Barbershops Completing all Components of CLIP | Month 12
  Measurement of the rate of adoption of Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP).
Number of Barbershops Continuing to Use CLIP at 6 Months Post-Completion of Intervention | Month 18
  Measurement of the sustainability of Community-to-Clinic Linkage Implementation Program in Barbershops (CLIP).
Number of Participants Presenting with Incident Stage 2 HTN | Baseline
  Incident Stage 2 hypertension (HTN) is defined as:
  * Systolic Blood Pressure (SBP) of at least 140 millimeters of mercury (mm Hg)/Diastolic Blood Pressure (DBP) of at least 90 mm Hg; or
  * Antihypertensive medication initiation.
Number of Participants Presenting with Incident Stage 2 HTN | Month 6
  Incident Stage 2 hypertension (HTN) is defined as:
  * Systolic Blood Pressure (SBP) of at least 140 millimeters of mercury (mm Hg)/Diastolic Blood Pressure (DBP) of at least 90 mm Hg; or
  * Antihypertensive medication initiation.
Number of Participants Presenting with Incident Stage 2 HTN | Month 12
  Incident Stage 2 hypertension (HTN) is defined as:
  * Systolic Blood Pressure (SBP) of at least 140 millimeters of mercury (mm Hg)/Diastolic Blood Pressure (DBP) of at least 90 mm Hg; or
  * Antihypertensive medication initiation.
Number of Participants Presenting with Incident Stage 2 HTN | Month 18
  Incident Stage 2 hypertension (HTN) is defined as:
  * Systolic Blood Pressure (SBP) of at least 140 millimeters of mercury (mm Hg)/Diastolic Blood Pressure (DBP) of at least 90 mm Hg; or
  * Antihypertensive medication initiation.
12-Item Short Form Survey (SF-12) Questionnaire Score | Baseline
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the better the physical and mental health functioning.
12-Item Short Form Survey (SF-12) Questionnaire Score | Month 6
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the better the physical and mental health functioning.
12-Item Short Form Survey (SF-12) Questionnaire Score | Month 12
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the better the physical and mental health functioning.
12-Item Short Form Survey (SF-12) Questionnaire Score | Month 18
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality-of-life measure. SF-12 consists of 12 questions that are scored in various ways. The total score range is 12-48; the higher the score, the better the physical and mental health functioning.
Cost per Millimeters of Mercury (mm Hg) Reduction in Blood Pressure (BP) | Up to Month 18
  Dollar amount associated with a 1-mm Hg reduction in BP. Lower costs are considered more desirable outcomes.
Cost per Incident Stage 2 Hypertension (HTN) Case Prevented | Up to Month 18
  Dollar amount associated with the prevention of an Incident Stage 2 HTN case. Lower costs are considered more desirable outcomes.
  Incident Stage 2 HTN is defined as:
  * Systolic Blood Pressure (SBP) of at least 140 millimeters of mercury (mm Hg)/Diastolic Blood Pressure (DBP) of at least 90 mm Hg; or
  * Antihypertensive medication initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ravenell, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to:
  Joseph Ravenell, MD Telephone: 646-501-9932 Email: Joseph.Ravenell@nyulangone.org
  The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access upon reasonable request. Requests should be directed to Joseph.Ravenell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Arabadjian M, Green T, Foti K, Dubal M, Poudel B, Christenson A, Wang Z, Dietz K, Brown D, Liriano K, Onaga E, Mantello G, Schoenthaler A, Cooper LA, Spruill TM, Ogedegbe G, Ravenell J. Community Engagement for Effective Recruitment of Black Men at Risk for Hypertension: Baseline Data From the Community-to-Clinic Program (CLIP) Randomized Controlled Trial. Am J Hypertens. 2025 Oct 14;38(11):888-895. doi: 10.1093/ajh/hpaf099. PMID 40482027
- [Derived] Ravenell J, Green T, Arabadjian M, Schoenthaler A, Ogedegbe O. Barbershop-Facilitated Community-to-Clinic Linkage Implementation Program: Rationale and Protocol for a Novel Program to Prevent Hypertension Among Black Men. Am J Hypertens. 2023 Apr 15;36(5):240-247. doi: 10.1093/ajh/hpac133. PMID 37061797